CLINICAL TRIAL: NCT04710303
Title: Phase 1b Open-Label Study of the Safety, Reactogenicity, and Immunogenicity of a Prophylactic COVID-19 Vaccination Using a 2nd Generation (E1/E2B/E3-Deleted) Adenoviral Platform in Healthy South African Adults (ProVIVA-SA-1)
Brief Title: COVID-19 Vaccination Using a 2nd Generation (E1/E2B/E3-Deleted) Adenoviral Platform in Healthy South African Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AW_001_ProVIVA-SA-1
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) per dose (Experimental): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) per dose on Days 1 and 22
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 2 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP per dose (Experimental): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP per dose on Days 1 and 22
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP per dose (Experimental): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP per dose (or 5 × 10e10 VP per dose if safety concerns identified at higher dose) on Day 1
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP per dose (Experimental): hAd5-S-Fusion+N-ETSD at 2 × 10e10 VP per nostril (or 4 × 10e10 VP per dose) on Day 1
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine

INTERVENTIONS:
Biological: hAd5-S-Fusion+N-ETSD vaccine — The hAd5-S-Fusion+N-ETSD vaccine is a hAd5 [E1-, E2b-, E3-] vector-based targeting vaccine encoding the SARS-CoV-2 S and N proteins. The hAd5-S-Fusion+N-ETSD vaccine is designed to induce both humoral and cellular responses even in individuals with pre-existing adenoviral immunity.

SUMMARY:
This is a phase 1b, open-label study in adult healthy participants. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of the hAd5-S-Fusion+N-ETSD vaccine and select a dose for future studies.

ELIGIBILITY:
Inclusion Criteria

1. Adults, age 18 - 50 years, inclusive, at time of first study vaccination.
2. Able to understand and provide a signed informed consent that fulfils the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
3. Agrees to the collection of biospecimens (e.g. nasopharyngeal [NP] swabs) and venous blood per protocol.
4. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
5. Body mass index (BMI) < 30.00 kg/m2
6. Temperature < 38.0°C on day of first study vaccination.
7. Good general health as shown by medical history, physical exam, and screening laboratory tests
8. Screen negative for Tuberculosis per local screening guidelines
9. Male participants should all be at low risk of HIV acquisition based on pre-specified, validated criteria(Laher 2014) i.e. answering YES to any of the following questions:

1. Are you sexually abstinent? 2. Are you in a mutually monogamous relationship with a known HIV-uninfected partner? 3. Have you had only one partner in the preceding 12 months who is believed to be HIV-uninfected and with whom condoms were used regularly?

Laboratory Inclusion Values/ Results:

10. Alanine aminotransferase (ALT) <1.1 times the upper limit of normal 11. Serum Creatinine <80 umol/L in females and <106 umol/L in males 12. Haemoglobin >12.0g/dL in females and >13.5g/dL in males 13. Platelets >150 x 109/L in all participants 14. No serological evidence of chronic infection with Hepatitis B (hepatitis B surface antigen (HepBSAg) negative by a locally approved assay) done during the screening period 15. No serological evidence of chronic infection with Hepatitis C (hepatitis C antibody(anti-HCV) negative by a locally approved assay) done during the screening period 16. Negative for SARS-CoV-2 (qPCR test) on NP swab(or other appropriate respiratory specimen) within 3 days prior to the first study vaccination 17. No serological evidence of prior infection with SARS-CoV-2 (by a locally approved assay) done during the screening period 18. A negative serum or urine pregnancy test during screening and on the day of and prior to each dose must be documented before the vaccine is administered to a female participant.

19. Negative for HIV-1 and -2 on blood test(by either 2 rapid tests or an ELISA, both must be locally approved assays) done during the screening period.

Reproductive Status:

20. Female participants of childbearing potential must agree to use effective contraception for sexual activity that may lead to pregnancy while on study until at least 30 days after the last dose of the study vaccine. Effective contraception for female participants includes:

* Intrauterine device (IUD), or
* Hormonal contraception (oral/ injectable/ implant/ transdermal etc.) Or; 21. Non-sterile male participants must agree to use a condom while on study until at least 30 days after the last dose of the study vaccine.

Or; 22. Participant must not be of reproductive potential or sterile(as verified by medical records), such as:

* Having been diagnosed with menopause(with no menses for 1 year)
* Having undergone hysterectomy, bilateral oophorectomy or orchidectomy
* Having undergone surgical sterilization (e.g., vasectomy, tubal ligation)

Exclusion Criteria:

1. A history of illness compatible with COVID-19 disease since March 2020.
2. Serious adverse reaction to any vaccine, any unrelated medication or any component of the investigational vaccine, including a history of anaphylaxis and symptoms of a severe allergic reaction and history of allergies in the past.
3. Pregnant or breastfeeding women.
4. Live in a nursing home or long-term care facility.
5. Chronic lung disease or moderate to severe asthma.
6. Bone marrow or organ transplantation recipients.
7. Diabetes.
8. Chronic kidney disease undergoing dialysis.
9. Liver disease.
10. Any disease associated with acute fever, or any infection.
11. Self-reported history of severe acute respiratory syndrome (SARS).
12. Chronic hepatitis B or hepatitis C infection.
13. HIV positive or other acquired or hereditary immunodeficiency.
14. Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension without controllable drugs, etc.
15. History of hereditary, idiopathic or acquired angioedema.
16. Urticaria in the last 12 months prior to screening.
17. No spleen or functional asplenia.
18. Platelet disorder or other bleeding disorder that may cause injection contraindication.
19. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness. (Including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators. The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.)
20. Prior administration of blood products within 120 days before first study vaccination.
21. Prior administration of other research medicines or investigational product within 30 days before first study vaccination.
22. Prior administration of attenuated vaccine within 30 days before first study vaccination..
23. Prior administration of inactivated vaccine within 14 days before first study vaccination.
24. Current treatment with investigational agents for prophylaxis of COVID-19.
25. Have a household contact that has been diagnosed with COVID-19 within 14 days before fist study vaccine.
26. Current anti-tuberculosis prophylaxis or therapy.
27. Currently receiving treatment for cancer or history of cancer in the last five years (except basal cell carcinoma of the skin and cervical carcinoma in situ).
28. According to the judgement of investigator any medical, psychiatric, psychological, social, occupational or other conditions that could affect the participants ability to sign informed consent, provide safety assessment data or comply with the requirements of the study protocol.
29. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Khayelitsha Clinical Research Site, Khayelitsha, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose: hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP per dose on Days 1 and 22
  hAd5-S-Fusion+N-ETSD vaccine: The hAd5-S-Fusion+N-ETSD vaccine is a hAd5 [E1-, E2b-, E3-] vector-based targeting vaccine encoding the SARS-CoV-2 S and N proteins. The hAd5-S-Fusion+N-ETSD vaccine is designed to induce both humoral and cellular responses even in individuals with pre-existing adenoviral immunity.
Period: Overall Study
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Started | 10 | 11 | 10 | 10
Completed | 10 | 7 | 10 | 10
Not Completed | 0 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose | Total
Number analyzed (Participants) | 10 | 11 | 10 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (7.88) | 28.4 (9.45) | 24.3 (5.46) | 22.1 (4.72) | 25.5 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 7 | 7 | 25
  Male | 4 | 6 | 3 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 11 | 10 | 10 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 11 | 10 | 10 | 40
  White | 1 | 0 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Cohorts 1 and 2 SARS-CoV-2 seronegative healthy volunteers [Count of Participants; unit: Participants] | 10 | 11 | 0 | 0 | 21
Cohorts 3 and 6 SARS-CoV-2 seropositive healthy volunteers [Count of Participants; unit: Participants] | 0 | 0 | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAE)
Description: Number of Participants with MAAEs through 1 week post final vaccine administration
Time Frame: From first dose of study treatment through 1 week post final vaccine administration; up to 29 days for Cohorts 1 and 2, and up to 8 days for Cohorts 3 and 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Solicited Local Reactogenicity AEs
Description: Number of Participants with solicited local reactogenicity AEs through 1 week post final vaccine administration
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 9 | 5 | 7 | 2

3. Primary Outcome: Number of Participants With Solicited Systemic Reactogenicity AEs
Description: Number of Participants with solicited systemic reactogenicity AEs through 1 week post final vaccine administration
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 6 | 5 | 6 | 4

4. Primary Outcome: Number of Participants With Unsolicited AEs
Description: Number of Participants with unsolicited AEs through 1 week post final vaccine administration
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 3 | 4 | 2 | 4

5. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAE)
Description: Number of Participants with MAAEs through 30 days post final vaccine administration
Time Frame: From first dose of study treatment through 30 days post final vaccine administration; up to 52 days for Cohorts 1 and 2 and up to 31 days for Cohorts 3 and 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 1 | 3 | 1 | 2

6. Primary Outcome: Number of Participants With Unsolicited AEs
Description: Number of Participants with unsolicited AEs through 30 days post final vaccine administration
Time Frame: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 4 | 7 | 3 | 5

7. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAE)
Description: Number of Participants with MAAEs through 6 months post final vaccine administration
Time Frame: From first dose of study treatment through 6 months post final vaccine administration; up to 202 days for Cohorts 1 and 2, and up to 181 days for Cohorts 3 and 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 2 | 3 | 2 | 4

8. Primary Outcome: Number of Participants With Unsolicited AEs
Description: Number of Participants with unsolicited AEs through 6 months post final vaccine administration
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (n = 10): hAd5-S-Fusion+N-ETSD at 5 × 10e10 Viral Particles (VP) Per Dose | Cohort 2 (n = 11): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 3 (n = 10): hAd5-S-Fusion+N-ETSD at 1 × 10e11 VP Per Dose | Cohort 6 (n=10):hAd5-S-Fusion+N-ETSD at 4 × 10e10 VP Per Dose
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 5 | 9 | 4 | 6

ADVERSE EVENTS:
Time Frame: Solicited AEs: From first dose to 1 week post final vaccine; up to 29 days for Cohorts 1 and 2, and up to 8 days for Cohorts 3 and 6. Unsolicited AEs: From first dose to 30 days post final vaccine; up to 52 days for Cohorts 1 and 2 and up to 31 days for Cohorts 3 and 6. Medically Attended AEs and Serious AEs: From first dose to 6 months post final vaccine; up to 202 days for Cohorts 1 and 2, and up to 181 days for Cohorts 3 and 6. SAEs related to treatment were reported any time, up to 1 year.
Groups:
- Group 1: Cohort 1; Group 1: Cohort 2; Group 1: Cohort 3; Group 1: Cohort 6: Incidence of Solicited Local Reactogenicity Adverse Events Through 1 Week Post Final Vaccine Administration
- Group 2: Cohort 1; Group 2: Cohort 2; Group 2: Cohort 3; Group 2: Cohort 6: Incidence of Solicited Systemic Reactogenicity Adverse Events Through 1 Week Post Final Vaccine Administration
- Group 3: Cohort 1; Group 3: Cohort 2; Group 3: Cohort 3; Group 3: Cohort 6: Incidence of Unsolicited Adverse Events Through 6 Months Post Final Vaccine Administration
- Group 4: Cohort 1; Group 4: Cohort 2; Group 4: Cohort 3; Group 4: Cohort 6: Incidence of Medically Attended Adverse Events Through 6 Months Post Final Vaccine Administration
Arm/Group | Group 1: Cohort 1 | Group 1: Cohort 2 | Group 1: Cohort 3 | Group 1: Cohort 6 | Group 2: Cohort 1 | Group 2: Cohort 2 | Group 2: Cohort 3 | Group 2: Cohort 6 | Group 3: Cohort 1 | Group 3: Cohort 2 | Group 3: Cohort 3 | Group 3: Cohort 6 | Group 4: Cohort 1 | Group 4: Cohort 2 | Group 4: Cohort 3 | Group 4: Cohort 6
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 5/11 | 7/10 | 2/10 | 6/10 | 5/11 | 6/10 | 4/10 | 5/10 | 9/11 | 4/10 | 6/10 | 2/10 | 3/11 | 2/10 | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Cohort 1 (N=10) | Group 1: Cohort 2 (N=11) | Group 1: Cohort 3 (N=10) | Group 1: Cohort 6 (N=10) | Group 2: Cohort 1 (N=10) | Group 2: Cohort 2 (N=11) | Group 2: Cohort 3 (N=10) | Group 2: Cohort 6 (N=10) | Group 3: Cohort 1 (N=10) | Group 3: Cohort 2 (N=11) | Group 3: Cohort 3 (N=10) | Group 3: Cohort 6 (N=10) | Group 4: Cohort 1 (N=10) | Group 4: Cohort 2 (N=11) | Group 4: Cohort 3 (N=10) | Group 4: Cohort 6 (N=10)
Injection site pruritus (General disorders) | 4 | 5 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 5 | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 6 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
HIV infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Cohort 4 (sublingual 1x10e11 VP per dose on Day 1) and Cohort 5 (sublingual and subcutaneous 1x10e11 VP for each dose on Day 1) did not enroll any subjects.

Only one AE table per AE category was presented to reduce data entry redundancy.

Only safety data is provided due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT04710303/Prot_SAP_000.pdf